CLINICAL TRIAL: NCT02819141
Title: Efficacy of Self-management of Sedative Therapy by Ventilated ICU Patients
Brief Title: Self-management of Sedative Therapy by Ventilated Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Minnesota (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Linda L. Chlan, Ph.D., R.N., FAAN, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-000417; 5R01HL130881 (NIH)
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Critical Illness; Anxiety; Respiratory Failure
MeSH Terms: conditions — Critical Illness; Anxiety Disorders; Respiratory Insufficiency | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): These patient will get usual care - sedation administered by ICU Nurses as deemed necessary by primary care team
- Dexmedetomidine (Experimental): These patients will receive a basal intravenous infusion of medication (Dexmedetomidine) and have access to self-administered sedation medication (Dexmedetomidine) for anxiety.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patient will receive a maintenance intravenous infusion of medication (Dexmedetomidine) and have access to self-controlled sedation medication (Dexmedetomidine) for anxiety.
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
The purpose of this randomized clinical trial is to test the efficacy of dexmedetomidine for the self-management of sedative therapy (SMST) in a sample of critically ill patients receiving mechanical ventilator support. The investigators hypothesis is that self-management of sedative therapy by mechanically ventilated patients in the intensive care unit (ICU), tailored to their individual needs will be more efficacious than nurse-administered sedative therapy in reducing anxiety, which may reduce duration of mechanical ventilator support and occurrence of delirium.

DETAILED DESCRIPTION:
The overall objective of this study is to demonstrate efficacy for conducting a future, pragmatic effectiveness trial to test whether self-management of sedative therapy (SMST) is superior to nurse-administered sedative therapy in day-to-day intensive care unit (ICU) practice. This efficacy trial is powered for the investigators primary, clinically relevant endpoints (anxiety, duration of mechanical ventilation, and delirium presence), and examines patient outcomes adversely affected by sedative administration practices, such as prolonged ICU stays, altered mental status, and diminished post-ICU quality of life. This randomized clinical trial with a total of 190 mechanically ventilated patients enrolled and maintained on protocol will address the following Specific Aims.

The primary aim is to determine the efficacy of SMST compared to nurse-administered sedative therapy on anxiety, duration of mechanical ventilation, and presence of delirium in mechanically ventilated patients (MVPs).

The secondary aim is to compare level of arousal and sedative exposure in mechanically ventilated patients (MVPs) randomized to SMST to those MVPs receiving nurse-administered sedative therapy. The investigators hypothesize that SMST patients will be easily arousable, more alert, and exposed to less sedation than those who receive nurse-administered sedative therapy.

Exploratory aims are to compare post-ICU outcomes (physical/functional status, psychological well-being, and health-related quality of life) and recall of ICU experiences between MVPs randomized to SMST and those receiving nurse-administered sedative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is acutely mechanically ventilated during the current hospitalization.
2. Subject is currently receiving a continuous intravenous infusion of a sedative/opioid medication(s) or has received at least one intravenous bolus dose of a sedative/opioid medication in the previous 24 hours (fentanyl, hydromorphone, ketamine, morphine, midazolam, diazepam, lorazepam, propofol, haloperidol, dexmedetomidine).
3. Subject must pass pre-Patient-Controlled Sedation (PCS) screening test and be assessed Richmond Agitation-Sedation Scale (RASS) -2 to +1
4. Subject Age ≥ 18 years
5. Subject or their proxy is capable of providing informed consent

Exclusion Criteria:

1. Aggressive ventilatory support or prone ventilation.
2. Hypotension (systolic blood pressure < 85 mmHg) requiring a vasopressor at a dose greater than norepinephrine or epinephrine 0.15 mcg/kg/min or vasopressin > 2.4 units per hour. Subjects will be excluded if they require more than one continuous infusion of a catecholamine vasopressor medication simultaneously. Subjects will be excluded if the vasopressor dose was higher than norepinephrine or epinephrine 0.15 mcg/kg/min, vasopressin > 2.4 units per hour, phenylephrine >3 mcg/kg/min, dopamine >10 mcg/kg/min or dobutamine at any dose in the prior 6 hours. If dopamine is being used to increase heart rate, rather than as a vasopressor for hypotension, subject will be excluded.
3. Second or third degree heart block or bradycardia (heart rate < 50 beats/min).
4. Paralysis or other condition preventing the use of push button device
5. Positive pregnancy test or lactation
6. Acute hepatitis or liver failure (direct bilirubin >5 mg/dL)
7. Acute stroke or uncontrolled seizures.
8. Acute myocardial infarction within 48 hours prior to enrollment.
9. Severe cognition or communication problems (such as coma, deafness without signing literacy, physician-documented dementia)
10. Assessed RASS -3, -4, -5 or RASS +2,+3, +4
11. Chronic ventilator support in place of residence prior to current hospitalization.
12. Imminent extubation from mechanical ventilator support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2024-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Chlan, RN, PhD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - School of Medicine, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tracy MF, Chlan L, Savik K, Skaar DJ, Weinert C. A Novel Research Method for Determining Sedative Exposure in Critically Ill Patients. Nurs Res. 2019 Jan/Feb;68(1):73-79. doi: 10.1097/NNR.0000000000000322. PMID 30540694
- [Background] Chlan LL, Weinert CR, Tracy MF, Skaar DJ, Gajic O, Ask J, Mandrekar J. Study protocol to test the efficacy of self-administration of dexmedetomidine sedative therapy on anxiety, delirium, and ventilator days in critically ill mechanically ventilated patients: an open-label randomized clinical trial. Trials. 2022 May 16;23(1):406. doi: 10.1186/s13063-022-06391-w. PMID 35578315
- [Background] Chlan LL, Tracy MF, Ask J, Lal A, Mandrekar J. The impact of the COVID-19 pandemic on ICU clinical trials: a description of one research team's experience. Trials. 2023 May 11;24(1):321. doi: 10.1186/s13063-023-07355-4. PMID 37165383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Dexmedetomidine
Started | 81 | 80
Completed | 75 | 60
Not Completed | 6 | 20
Not completed — Extubated or discontinued prior to day 7 | 6 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Dexmedetomidine | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (13.8) | 56.2 (16.0) | 58.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 35 | 73
  Male | 43 | 45 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 81 | 79 | 160
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 5 | 7
  White | 75 | 74 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 81 | 80 | 161
Acute Physiology and Chronic Health Evaluation (APACHE) III score [Median (Inter-Quartile Range); unit: units on a scale] — APACHE III is a measure of illness severity and prognostication of hospital mortality for critically ill patients admitted to the intensive care unit. Scores range from 0 to 299 with higher scores indicating more ill and associated with an increased risk of death. APACHE III scores are calculated based on the worst value within the first 24 hours of ICU admission including temperature, blood pressure, heart rate, oxygenation, pH, kidney function, blood counts, neurological status, age, chronic health conditions.
  units on a scale | 80.0 [63 to 101] | 85.5 [58.5 to 104.5] | 82 [60 to 102]

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Rating Using the 100mm Vertical Visual Analog Scale
Description: Vertical visual analog scale will be used to measure level of state anxiety from 0/zero (no anxiety) to 100 (most anxiety ever). Higher scores mean more anxiety.
Time Frame: 7 days
Population: Not all enrolled patients able to respond to each assessment time point for anxiety ratings. They may have been extubated and completed the ICU study phase, withdrew from the study, or died.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dexmedetomidine: These patients will receive a basal intravenous infusion of medication (Dexmedetomidine) and have access to self-administered sedation medication (Dexmedetomidine) for anxiety.
  Dexmedetomidine: Patient will receive a basal intravenous infusion of medication (dexmedetomidine) and have access to self-administered bolus doses of dexmedetomidine for anxiety.
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
score on a scale
  Day 1 morning: number analyzed (Participants) | 51 | 50
  Day 1 morning | 44.4 (33.2) | 43.4 (33.4)
  Day 1 afternoon: number analyzed (Participants) | 42 | 37
  Day 1 afternoon | 40.5 (31.8) | 33.1 (30.9)
  Day 1 evening: number analyzed (Participants) | 30 | 26
  Day 1 evening | 45.1 (32.4) | 40.9 (35.7)
  Day 2 morning: number analyzed (Participants) | 33 | 25
  Day 2 morning | 49.8 (30.9) | 44.6 (34.4)
  Day 2 afternoon: number analyzed (Participants) | 28 | 20
  Day 2 afternoon | 41.9 (33.4) | 41.4 (38.5)
  Day 2 evening: number analyzed (Participants) | 22 | 16
  Day 2 evening | 50.9 (32.7) | 54.9 (36.3)
  Day 3 morning: number analyzed (Participants) | 26 | 19
  Day 3 morning | 48 (35.0) | 49.8 (39.8)
  Day 3 afternoon: number analyzed (Participants) | 20 | 13
  Day 3 afternoon | 43.3 (33.9) | 58.6 (40.1)
  Day 3 evening: number analyzed (Participants) | 21 | 8
  Day 3 evening | 47.3 (39.2) | 48.1 (33.1)
  Day 4 morning: number analyzed (Participants) | 17 | 8
  Day 4 morning | 43.4 (35.0) | 52.4 (30.8)
  Day 4 afternoon: number analyzed (Participants) | 20 | 10
  Day 4 afternoon | 43.3 (35.5) | 51.4 (36.9)
  Day 4 evening: number analyzed (Participants) | 16 | 9
  Day 4 evening | 48.2 (34.7) | 44.1 (39.7)
  Day 5 morning: number analyzed (Participants) | 16 | 8
  Day 5 morning | 49.1 (31.6) | 36.1 (32.3)
  Day 5 afternoon: number analyzed (Participants) | 16 | 8
  Day 5 afternoon | 39.6 (27.4) | 32.0 (28.7)
  Day 5 evening: number analyzed (Participants) | 13 | 8
  Day 5 evening | 50.7 (37.6) | 39.6 (25.6)
  Day 6 morning: number analyzed (Participants) | 15 | 7
  Day 6 morning | 39.5 (31.1) | 46.1 (31.4)
  Day 6 afternoon: number analyzed (Participants) | 12 | 6
  Day 6 afternoon | 33.1 (28.0) | 53.3 (26.9)
  Day 6 evening: number analyzed (Participants) | 12 | 5
  Day 6 evening | 55.7 (33.1) | 38.0 (34.4)
  Day 7 morning: number analyzed (Participants) | 11 | 5
  Day 7 morning | 47.0 (29.3) | 74.4 (14.9)
  Day 7 afternoon: number analyzed (Participants) | 5 | 4
  Day 7 afternoon | 34.4 (35.8) | 30.8 (14.8)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; We estimated the power for multilevel models approximating our study design. A sample size of 95 patients per arm, 190 total (at a minimum 7 data collection points for each, resulting in ~1,050 observations) will have greater than 80% power to detect small to moderate effects (i.e., 0.11 or greater) in between-group differences in anxiety, delirium, and duration of mechanical ventilation at alpha = .05 for all proposed models; Test type: Superiority; p = 0.30, Generalized estimating equations — A priori threshold for statistical significance was p < 0.05; Controlling for age, daily sequential organ failure assessment (SOFA) score, sedation intensity, and time of day of assessment
Statistical Analysis 2: Comparison: Control vs Dexmedetomidine; Test type: Superiority — Controlling for time of day, study day, age, sex, illness severity, and sedation frequency; p = 0.9858, Generalized Estimating equations

2. Primary Outcome: Duration of Mechanical Ventilatory Support After Study Enrollment
Description: Duration of time (hours) patients received mechanical ventilatory support after randomization to either Control or dexmedetomidine self-management of sedative therapy to extubation.
Time Frame: 7 days
Population: Includes all patients enrolled who were randomized using an Intention to treat analysis
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
hours | 68.7 (58.2) | 50.3 (52.8)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.02, t-test, 1 sided — a priori threshold for significance p < 0.05

3. Primary Outcome: Incidence of Delirium Using the Confusion Assessment Method-ICU (CAM-ICU)
Description: Confusion Assessment Method-ICU (CAM-ICU) used to assess for the presence (CAM-ICU+) or absence (CAM-ICU-) of delirium at each assessment.
Time Frame: 7 days
Measure: Number; unit: participants CAM-ICU+
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
participants CAM-ICU+
  Study entry CAM-ICU+ | 15 | 7
  Day #1 CAM-ICU+ | 14 | 10
  Day #2 CAM-ICU+ | 9 | 5
  Day #3 CAM-ICU+ | 8 | 3
  Day #4 CAM-ICU+ | 2 | 2
  Day #5 CAM-ICU+ | 2 | 2
  Day #6 CAM-ICU+ | 0 | 4
  Day #7 CAM-ICU+ | 0 | 2
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.97, Generalized estimating equations; Controlling for sedation intensity, age, daily Sequential Organ Failure Assessment (SOFA) score, study day, and time of day assessment
Statistical Analysis 2: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.5647, Generalized estimating equations; Controlling for sedation frequency, age, sex, illness severity, study day, and time of day assessment

4. Secondary Outcome: Comparison of Level of Arousal and Agitation Using the Richmond Agitation-Sedation Scale (RASS)
Description: The Richmond Agitation-Sedation Scale (RASS) was used to assess the level of alertness and agitation in enrolled patients. Scores range from -5 to +4. RASS 0/zero indicates alert and calm patient. Negative scores (-1 to -5) indicate increasing level of sedation with -5 indicating unarousable. Positive scores indicate increasing agitation (+1 to +4) with +4 indicating a combative patient. For enrolled study patients, RASS score -2 (light sedation) to +1 (restless) was considered in range. We report here the total number of patients assessed as outside the desirable range of RASS score -5 to -3 and +2 to +4 by each ICU study day.
Time Frame: 7 days
Population: Not all patients were available for RASS assessment at each time point as some patients were extubated and completed the study, or were withdrawn or died.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
Participants
  Day #1 : Number of patients assessed: number analyzed (Participants) | 65 | 68
  Day #1 : Number of patients assessed | 65 | 68
  Day #1 : Number of patients out of range: number analyzed (Participants) | 65 | 68
  Day #1 : Number of patients out of range | 12 | 5
  Day #2 : Number of patients assessed: number analyzed (Participants) | 42 | 32
  Day #2 : Number of patients assessed | 42 | 32
  Day #2 : Number of patients out of range: number analyzed (Participants) | 42 | 32
  Day #2 : Number of patients out of range | 7 | 5
  Day #3 : Number of patients assessed: number analyzed (Participants) | 36 | 22
  Day #3 : Number of patients assessed | 36 | 22
  Day #3 : Number of patients out of range: number analyzed (Participants) | 36 | 22
  Day #3 : Number of patients out of range | 6 | 3
  Day #4 : Number of patients assessed: number analyzed (Participants) | 27 | 12
  Day #4 : Number of patients assessed | 27 | 12
  Day #4 : Number of patients out of range: number analyzed (Participants) | 27 | 12
  Day #4 : Number of patients out of range | 2 | 4
  Day #5 : Number of patients assessed: number analyzed (Participants) | 20 | 12
  Day #5 : Number of patients assessed | 20 | 12
  Day #5 : Number of patients out of range: number analyzed (Participants) | 20 | 12
  Day #5 : Number of patients out of range | 2 | 3
  Day #6 : Number of patients assessed: number analyzed (Participants) | 17 | 10
  Day #6 : Number of patients assessed | 17 | 10
  Day #6 : Number of patients out of range: number analyzed (Participants) | 17 | 10
  Day #6 : Number of patients out of range | 1 | 3
  Day #7 : Number of patients assessed: number analyzed (Participants) | 14 | 20
  Day #7 : Number of patients assessed | 14 | 20
  Day #7 : Number of patients out of range: number analyzed (Participants) | 14 | 20
  Day #7 : Number of patients out of range | 1 | 1
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.39, Generalized estimating equation; controlling for age, daily Sequential Organ Failure Assessment (SOFA) score, time of day of assessment

5. Secondary Outcome: Comparison of Daily Sedation Intensity Each ICU Study Day Using Electronic Health Record Medication Data of Any of Nine Intravenous Sedative Medications Administered to Patients.
Description: Sedation intensity combines the number of sedative doses and the dose amount of any of 9 intravenous (IV) sedative medications (lorazepam, midazolam, propofol, morphine, hydromorphone, dexmedetomidine, fentanyl, haloperidol, ketamine) recorded in the electronic health record, summarized over all patients and time periods each day to obtain medians and quartiles. Each of the 9 sedative drugs administered during each 4-hr period is then assigned a ranking: 0 for drug not used, 1 for the bottom quartile, 2 for the second quartile, 3 for the third, and 4 for the fourth. A score is determined by summing for the 24-hr day over the 6, 4-hour blocks to produce a daily Sedation Intensity Score from 0-36, higher score more intense dosing received of sedative medications.
Time Frame: Daily Sedation intensity over a 7-day ICU study protocol period
Population: Patients exit the study at various times over the 7-day ICU study period leading to a different number of patients available for analysis on each ICU study day.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
score on a scale
  Study entry sedation intensity | 10.2 (6.6) | 9.1 (6.9)
  Day #1 sedation intensity: number analyzed (Participants) | 68 | 68
  Day #1 sedation intensity | 17.3 (12.0) | 16.6 (13.1)
  Day #2 sedation intensity: number analyzed (Participants) | 44 | 34
  Day #2 sedation intensity | 17.4 (13.0) | 20.7 (15.8)
  Day #3 sedation intensity: number analyzed (Participants) | 35 | 23
  Day #3 sedation intensity | 17.5 (14.2) | 19.8 (13.1)
  Day #4 sedation intensity: number analyzed (Participants) | 29 | 13
  Day #4 sedation intensity | 17.5 (13.3) | 24.2 (12.7)
  Day #5 sedation intensity: number analyzed (Participants) | 23 | 13
  Day #5 sedation intensity | 17.9 (15.2) | 25.7 (18.9)
  Day #6 sedation intensity: number analyzed (Participants) | 18 | 12
  Day #6 sedation intensity | 16.9 (18.8) | 22.8 (10.6)
  Day #7 sedation intensity: number analyzed (Participants) | 12 | 10
  Day #7 sedation intensity | 10.8 (13.8) | 13.5 (6.2)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.37, GEE

6. Other Pre Specified Outcome: Comparison of Post-ICU Physical Status Using the Katz Activities of Daily Living Scale
Description: Physical status will be assessed by the Katz Activities of Daily Living scale to assess basic physical abilities like bathing, feeding with 6 questions. Higher scores of 6 indicates the individual is independent, whereas a score of 0 indicates the individual is very dependent.
Time Frame: Independence in activities of daily living at 3 months and 6 months after hospital discharge over the telephone
Population: Different number of patients responded to the telephone call at each time point
  .
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 39 | 30
score on a scale
  3 months after discharge | 5.1 (1.8) | 5.6 (1.0)
  6 months after discharge: number analyzed (Participants) | 32 | 30
  6 months after discharge | 5.5 (1.2) | 5.6 (1.1)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.17, t-test, 1 sided
Statistical Analysis 2: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.81, t-test, 1 sided

7. Other Pre Specified Outcome: Comparison of Post-ICU Psychological Well-being Status Using the Patient Health Questionnaire-9
Description: Psychological well-being will be assessed by the Patient Health Questionnaire (PHQ-9) is a 9-item tool that tracks symptoms of major depression. Scores range from 9-36, with higher scores indicating altered psychological well-being.
Time Frame: 3 and 6 months after ICU discharge over the telephone
Population: 3 month PHQ-9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 36 | 28
score on a scale
  3 months after discharge | 23.0 (4.3) | 22.1 (5.2)
  6 months after discharge: number analyzed (Participants) | 30 | 28
  6 months after discharge | 23.5 (3.8) | 23.3 (4.1)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.47, t-test, 1 sided
Statistical Analysis 2: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.82, t-test, 1 sided

8. Other Pre Specified Outcome: Comparison of Post-ICU Psychological Well-being Status Using the Posttraumatic Stress Disorder Checklist Event Specific (PCL) Scale
Description: Psychological well-being will be assessed with the Posttraumatic Stress Disorder Checklist Event Specific (PCL) to measure symptoms of posttraumatic stress disorder after a stressful life experience of ICU admission. Scores range from 17-85 with higher scores indicating being symptomatic for posttraumatic stress.
Time Frame: 3 months and 6 months after ICU discharge over the telephone
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 38 | 30
score on a scale | 23.8 (7.4) | 27.7 (15.0)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; 3 months after ICU discharge; Test type: Superiority; p = 0.164, t-test, 1 sided
Statistical Analysis 2: Comparison: Control vs Dexmedetomidine; 6 months after ICU discharge; Test type: Superiority; p = 0.84, t-test, 1 sided

9. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Physical Function Domain
Description: Post-intensive care unit health-related quality of life will be assessed by the Short-Form-36 (SF-36) at 3- and 6-months after hospital discharge. The SF-36 tracks how well an individual feels and how well they are able to do their usual activities in eight health domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. A higher score defines a more favorable health state scored on a 0-100 range for each of the 8 domain scales.
Time Frame: 3 months after ICU discharge over the telephone Physical Function Domain
Population: Physical Function at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 30
score on a scale | 45.4 (29.9) | 53.8 (29.9)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.26, t-test, 1 sided

10. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Physical Function Domain
Description: Post-intensive care unit health-related quality of life will be assessed by the Short-Form-36 at 3- and 6-months after hospital discharge. The SF-36 tracks how well an individual feels and how well they are able to do their usual activities in eight health domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. A higher score defines a more favorable health state scored on a 0-100 range for each of the 8 domain scales.
Time Frame: 6 months after ICU discharge over the telephone Physical Function Domain
Population: Physical Function at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 57.0 (26.6) | 58.6 (30.7)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.82, t-test, 1 sided

11. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Role Limitations Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone Role Limitations Domain due to Physical Health
Population: Role limitations due to physical health at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 38 | 28
score on a scale | 22.4 (32.8) | 43.8 (38.9)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.018, t-test, 1 sided

12. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Role Limitations Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone Role Limitations Domain due to Physical Health
Population: Role limitations due to physical health at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 39.8 (38.0) | 44.2 (39.8)
Statistical Analysis 1: Comparison: Control; Test type: Superiority; p = 0.66, t-test, 1 sided

13. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Personal or Emotional Health Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone Role Limitations due to Personal or Emotional Health
Population: Role limitations due to personal or emotional health at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 80.2 (32.8) | 76.2 (33.8)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.63, t-test, 1 sided

14. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Using Personal or Emotional Health Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone Role Limitations due to Personal or Emotional Health
Population: Role limitations due to personal or emotional health at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 78.9 (34.4) | 71.4 (37.2)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.41, t-test, 1 sided

15. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Using the Energy/Fatigue Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone Energy/Fatigue Domain
Population: Energy/fatigue at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 54.3 (19.2) | 43.6 (26.7)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.06, t-test, 1 sided

16. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Using the Energy/Fatigue Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone Energy/Fatigue
Population: Energy/fatigue at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 54.2 (22.5) | 53.8 (20.2)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.93, t-test, 1 sided

17. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Emotional Well-being Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone Emotional Well-being
Population: Emotional well-being at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 83.5 (14.7) | 80.0 (21.1)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.43, t-test, 1 sided

18. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Emotional Well-being Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone Emotional Well-being
Population: Emotional well-being at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 81.8 (18.8) | 83.5 (15.5)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.69, t-test, 1 sided

19. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Social Functioning Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone social functioning
Population: Social functioning at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 76.4 (22.6) | 75.9 (27.8)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.94, t-test, 1 sided

20. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Socia Functioning Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone social functioning
Population: Social functioning at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 77.3 (24.3) | 72.5 (31.7)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.50, t-test, 1 sided

21. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Bodily Pain Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone bodily pain
Population: Bodily pain at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 72.3 (25.5) | 58.1 (27.7)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.03, t-test, 1 sided

22. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 Bodily Pain Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone bodily pain
Population: Bodily pain at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 71.0 (23.5) | 61.3 (31.6)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.17, t-test, 1 sided

23. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 General Health Domain
Description: as for outcome 10
Time Frame: 3 months after ICU discharge over the telephone general health perceptions
Population: General health perceptions at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 37 | 28
score on a scale | 52.3 (21.0) | 51.3 (24.2)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.85, t-test, 1 sided

24. Other Pre Specified Outcome: Comparison of Post-intensive Care Unit Health-related Quality of Life Using the Short-Form 36 General Health Domain
Description: as for outcome 10
Time Frame: 6 months after ICU discharge over the telephone general health perceptions
Population: General health perceptions at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 32 | 30
score on a scale | 52.7 (22.0) | 53.0 (26.9)
Statistical Analysis 1: Comparison: Control vs Dexmedetomidine; Test type: Superiority; p = 0.95, t-test, 1 sided

25. Secondary Outcome: Comparison of Daily Sedation Frequency Using Electronic Health Record Medication Data of Any of Nine Intravenous Sedative Medications Administered to Patients.
Description: Sedation Frequency is the number of individual intravenous (IV) sedative medication(s) doses administered to patients over each 24-hour day of lorazepam, midazolam, propofol, morphine, hydromorphone, dexmedetomidine, fentanyl, haloperidol, ketamine. Sedation frequency ranges from 0-216 with a higher number indicating more frequent receipt of a sedative medication(s).
Time Frame: Daily Sedation Frequency over a 7-day ICU study protocol period
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: count of sedative medication doses
Arm/Group | Control | Dexmedetomidine
Number analyzed (Participants) | 81 | 80
count of sedative medication doses
  Study entry sedation frequency | 13.9 (8.0) | 13.5 (7.3)
  Day #1 sedation frequency: number analyzed (Participants) | 68 | 68
  Day #1 sedation frequency | 24.6 (15.1) | 22.9 (13.5)
  Day #2 sedation frequency: number analyzed (Participants) | 44 | 34
  Day #2 sedation frequency | 24.3 (17.2) | 25.0 (15.5)
  Day #3 sedation frequency: number analyzed (Participants) | 35 | 23
  Day #3 sedation frequency | 24.4 (17.7) | 24.3 (14.1)
  Day #4 sedation frequency: number analyzed (Participants) | 29 | 13
  Day #4 sedation frequency | 25.0 (16.3) | 30.2 (14.8)
  Day #5 sedation frequency: number analyzed (Participants) | 23 | 13
  Day #5 sedation frequency | 25.9 (17.9) | 32.5 (19.0)
  Day #6 sedation frequency: number analyzed (Participants) | 18 | 12
  Day #6 sedation frequency | 23.5 (19.3) | 27.3 (10.9)
  Day #7 Sedation frequency: number analyzed (Participants) | 12 | 10
  Day #7 Sedation frequency | 14.9 (14.2) | 16.0 (10.2)

ADVERSE EVENTS:
Time Frame: Adverse Event Data were collected from study enrollment day 0 to day 7 of the ICU phase plus an additional 24 hours after completion of the 7-day ICU phase for a total maximum of 8 days.
Arm/Group | Control | Dexmedetomidine
All-Cause Mortality (participants affected / at risk) | 1/81 | 0/80
Serious Adverse Events (participants affected / at risk) | 5/81 | 12/80
Other Adverse Events (participants affected / at risk) | 29/81 | 24/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=81) | Dexmedetomidine (N=80)
Worsening respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) — Worsening respiratory failure with increasing sedation needs
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) — Cardiac arrest
Device disruption (General disorders) | 3 (3) | 2 (2) — Self-removal of endotracheal tube or dislodged feeding tube or ventilator tubing
Persistent agitation (General disorders) | 0 (0) | 3 (3) — Persistent anxiety or agitation
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=81) | Dexmedetomidine (N=80)
Hypotension (Cardiac disorders) | 23 (23) | 22 (22) — Hypotension
Bradycardia (Cardiac disorders) | 0 (0) | 2 (2) — Bradycardia
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) — Hypertension
Tachycardia (Cardiac disorders) | 5 (5) | 0 (0) — Tachycardia

LIMITATIONS AND CAVEATS:
The corona virus (COVID-19) global pandemic adversely impacted the ICU clinical trial. The pandemic influenced many aspects of patient availability for enrollment, changes to patient management including sedation regimens and clinical practice in the care of critically ill patients receiving mechanical ventilatory support. Fewer than planned patients randomized to dexmedetomidine self-management of sedative therapy actually received the experimental intervention, resulting in unbalanced numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/41/NCT02819141/Prot_SAP_000.pdf
  • Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/41/NCT02819141/ICF_001.pdf